CLINICAL TRIAL: NCT04318977
Title: rTMS Add on Value for Amelioration of Negative Symptoms of Schizophrenia
Acronym: RADOVAN
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Regensburg (Other)
Collaborators: University Hospital, Aachen (Other); University Hospital Ostrava (Other); Brno University Hospital (Other)
Responsible Party: Principal Investigator, Berthold Langguth, MD, Ph.D., Clinical Professor, University of Regensburg
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 19-1616-101
Record Dates: First submitted 2020-03-16; First posted 2020-03-24 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Negative Symptoms With Primary Psychotic Disorder; Schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Intervention Model Description: randomized controlled trial with two active and one placebo arm
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- high-frequency repetitive transcranial magnetic stimulation (Experimental): repetitive transcranial magnetic stimulation over left dorsolateral prefrontal cortex using 3000 pulses applied with 10Hz and 120% resting motor threshold
  Interventions: Device: high-frequency rTMS
- theta burst stimulation (Experimental): intermittent theta burst stimulation over left dorsolateral prefrontal cortex using 600 pulses applied in trains of 10 triplets/bursts (50Hz) with 8s intertrain-interval and 120% resting motor threshold
  Interventions: Device: TBS
- sham rTMS (Placebo Comparator): half of the patients with high-frequency repetitive transcranial magnetic stimulation and half of the patients with theta burst Stimulation with angled coil (45 degree) or sham coil
  Interventions: Device: placebo

INTERVENTIONS:
Device: high-frequency rTMS — repetitive transcranial magnetic stimulation
  Arms: high-frequency repetitive transcranial magnetic stimulation
Device: TBS — theta burst stimulation
  Arms: theta burst stimulation
Device: placebo — placebo transcranial magnetic stimulation
  Arms: sham rTMS

SUMMARY:
Treatment of depression with repetitive transcranial magnetic stimulation (rTMS) has shown high evidence using high-frequency left dorsolateral prefrontal cortex (DLPFC) stimulation. The treatment of negative symptoms with the same protocol in schizophrenia is considered as possible effective. Theta burst stimulation is a new protocol which is characterized by shorter sessions showing first evidence that it's efficacy is comparable to the high-frequency rTMS. In this randomized placebo-controlled study the efficacy of high-frequency rTMS and TBS are evaluated.

DETAILED DESCRIPTION:
In this randomized placebo-controlled study the efficacy of high-frequency rTMS and TBS are evaluated. The active study arms are high-frequency rTMS and iTBS of the left dorsolateral prefrontal cortex to treat negative symptoms in schizophrenia. The control arm will include the same number of patients as each active arm and includes both sham rTMS and sham iTBS in the same proportion as the active treatments.

Standards of the trial will be harmonized across four clinical centers with the aim to pool data for analysis. Each center is responsible for ethical approval and adherence to good clinical practice by itself (Sponsor).

Interim analysis: Several meta-analyses of the effect of rTMS/iTBS on negative symptoms in schizophrenia showing heterogeneous effect sizes have been published since begin of the trial. Thefore, an interim analysis after inclusion of at least 15 patients in each arm was added to the protocol. In case of null findings and low effect sizes (no differences of either rTMS or TBS vs. sham in the primary outcome), the trial will be terminated.

ELIGIBILITY:
Inclusion Criteria:

* ICD-10: schizophrenia with primarily negative symptoms
* Age: 18-75 years
* at least 35 Points at the composite score of the SANS
* stabe medication during the last 2 weeks (at the investigator's discretion)
* written informed consent (by the patient or guardian)

Exclusion Criteria:

* clinically relevant unstable concomitant somatic diseases
* previous treatment by rTMS
* conditions in which TMS may not be applicated, as e.g., cardiac pacemakers or ferromagnetic implants
* history of epileptic seizures
* current substance or alcohol abuse, or clinically relevant comorbidity (according to M.I.N.I. interview)
* unacceptable concomitant medication (benzodiazepines in higher doses, e.g., Lorazepam > 2 mg/d, Diazepam > 10 mg/d)
* insufficient knowledge of the language of the country of the treatment site
* pregnancy and nursing period
* current statutory hospitalisation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2024-08-14 (Actual); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Scale for the Assessement of Negative Symptoms (SANS) | 4 weeks
  negative symptoms in schizophrenia with 25 items and a range 0-125 with higher score representing more symptoms

SECONDARY OUTCOMES:
Scale for the Assessement of Negative Symptoms (SANS) | 2 weeks, 4 weeks, 12 weeks
  negative symptoms in schizophrenia with 25 items and a range 0-125 with higher score representing more symptoms
Positive and Negative syndrome scale (PANSS) | 2 weeks, 4 weeks, 12 weeks
  positive and negative symptoms in schizophrenia with 30 items and a range 30-210 with higher scores representing more symptoms (total score, score for positive, negative symptoms and for general psychopathology)
Calgary Depression Scale for Schizophrenia (CDSS) | 2 weeks, 4 weeks, 12 weeks
  Calgary Depression Scale for Schizophrenia
Clinical global impression (CGI) | 2 weeks, 4 weeks, 12 weeks
  measure of overall symptom severity and treatment response on a scale 1-7 with higher scores presenting more symptoms
Major Depression Inventory (MDI) | 2 weeks, 4 weeks, 12 weeks
  measurment of depressivity: 10 items with a range 0-50 and higher values indicating higher scores
Hamilton depression rating scale (HDRS) | 2 weeks, 4 weeks, 12 weeks
  measurment of depressivity: 21 items with a range 0-65 and higher values indicating higher scores
Memory span test (digit span) | 4 weeks, 12 weeks
  test for short-term and working memory
test of attention (d2) | 4 weeks, 12 weeks
  test of attention for measurement of concentration
Resting state electroencephalogram (EEG) | 4 weeks
  measurement of resting state electrophysiologic activity as indicated by frequency analysis and rTMS-evoked activity
magnetic resonance imaging (MRI) | 4 weeks
  structural, anatomical, diffusion weighted magnetic resonance imaging
cigarettes | 4 weeks, 12 weeks
  number of smoked cigarettes per week

CONTACTS AND LOCATIONS:
Overall Officials: Berthold Langguth, MD, PhD, Study Chair — University of Regensburg
Locations (4):
- Czechia (2):
  - Brno University Hospital, Brno
  - University Hospital Ostrava, Ostrava
- Germany (2):
  - University Hospital Aachen, Aachen
  - University of Regensburg, Regensburg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hebel T, Langguth B, Schecklmann M, Schoisswohl S, Staudinger S, Schiller A, Ustohal L, Sverak T, Horky M, Kasparek T, Skront T, Hyza M, Poeppl TB, Riester ML, Schwemmer L, Zimmermann S, Sakreida K. Rationale and study design of a trial to assess rTMS add-on value for the amelioration of negative symptoms of schizophrenia (RADOVAN). Contemp Clin Trials Commun. 2022 Jan 20;26:100891. doi: 10.1016/j.conctc.2022.100891. eCollection 2022 Apr. PMID 35128142